CLINICAL TRIAL: NCT02739750
Title: Pioglitazone and Lumbar Bone Marrow Fat in Chronic Kidney Disease (CKD) Sub-study to Protocol Number 1308084213
Brief Title: Pioglitazone and Lumbar Bone Marrow Fat in Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Ranjani Moorthi, Assistant Professor, Division of Nephrology, Indiana University
Other Study IDs: Indiana U 1511993513
Record Dates: First submitted 2016-03-23; First posted 2016-04-15 (Estimated); Last update posted 2022-01-26 (Actual); Status verified 2022-01

CONDITIONS: Polycystic Kidney Diseases
MeSH Terms: conditions — Polycystic Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention — There is no intervention for this study. It is a MRS.

SUMMARY:
Chronic Kidney Disease (CKD) is associated with bone changes and very high fracture rates. A component of bone is marrow. Bone marrow fat is increased in patients with CKD compared to those in the normal population of the same age. It is not clear if there will be changes in the marrow fact content in those with CKD on Pioglitazone. In people with normal kidney function, thiazolidinedione group of drugs have had variable effects on bone marrow fat content, as measured by MRS. This is important as changes in marrow fat are likely related to changes in the bone in patients with chronic kidney disease.

DETAILED DESCRIPTION:
If patients consent to participate in the ancillary study of marrow fat changes with pioglitazone, those that are randomized to placebo or 15 mg pioglitazone for 12 months (per the criteria in the main study) will also undergo magnetic resonance spectroscopy (MRS) of the lumbar spine at L1, L2 and L3. MR spectroscopy of the lumbar spine (if they choose as this is ancillary study) will be performed 3 times over the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Included subjects will be those who consent to the study of Pioglitazone in ADPKD (Protocol number 1308084213). Therefore inclusion and exclusion criteria are the same as for that study. Subjects will NOT be offered participation in the bone marrow fat study till after they consent for the FDA approved study. Subjects who withdraw from the FDA approved study will be withdrawn from this protocol.

Inclusion/Exclusion Criteria for NCT#02697617

* Male or female ADPKD patients aged 18-55
* eGFR at or above ≥ 50 ml/min/1.73 m2 by 4 parameter MDRD or CKD-Epiformulas
* normal liver enzymes (ALT/AST)
* fasting blood glucose between 70 and120
* for female patients, a willingness to use double contraception to avoid pregnancy while in study
* able to give informed consent
* In the opinion of the investigator, high likelihood of progressive kidney disease

Exclusion Criteria:

* diabetes, defined as any of the following: fasting blood sugar > 130 times two, HgbA1C > 7, on any blood sugar lowering medication, or past diagnosis of diabetes not occurring during pregnancy
* uncontrolled hypertension, defined as systolic > 150, diastolic > 90 despite an attempt by physician to titrate medications
* history of impaired systolic function (ejection fraction < 50%) by previous ECHO or known ischemic cardiovascular disease
* findings suggestive of a kidney disease other than ADPKD
* systemic illness requiring immunosuppressive or anti-inflammatory agents
* congenital absence of a kidney or history of a total nephrectomy
* history of cyst reduction or partial nephrectomy
* history of renal cyst aspiration within the previous year
* History of bladder cancer, or gross hematuria
* inability to undergo MRI due to implantable devices or foreign objects that preclude MRI
* active renal transplant
* allergy or sensitivity to any of the components of the test materials
* institutionalized
* currently pregnant or plans to become pregnant during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: PKD subjects that consent to the FDA study, number 1308084213, will be approached for consenting for this bone marrow fat study.
  Subject must be enrolled in NCT#02697617
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
The percent change in the bone marrow lipid fraction averaged between L2, L3 and L4 at baseline to 12 months and 12 months to 24 months. | Baseline, 12 months, 24 months
  Subjects will undergo and MRI at Baseline, 12 months, and 24 months to measure bone marrow.

CONTACTS AND LOCATIONS:
Overall Officials: Ranjani Moorthi, MD, Principal Investigator — Faculty
Locations (1):
- University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No